CLINICAL TRIAL: NCT01307696
Title: Multicenter Prospective Clinical Registry To Evaluate The Safety And Efficacy Of A Self-Expanding Multi-Layered Partially Resorbable Absorbable Lightweight Polypropylene Mesh Device (Proceed Ventral Patch® Or Pvp®) For The Treatment Of Small And Medium Umbilical Ventral Hernias
Brief Title: Self-Expanding Multi-Layered Partially Resorbable Lightweight Polypropylene Mesh Device (Proceed Ventral Patch® Or Pvp®) For The Treatment of Small and Medium Umbilical Ventral Hernias
Status: Completed | Type: Observational
Sponsor: Algemeen Ziekenhuis Maria Middelares (Other)
Responsible Party: Principal Investigator, Jan Bontinck, Doctor, Algemeen Ziekenhuis Maria Middelares
Other Study IDs: MM
Record Dates: First submitted 2011-03-02; First posted 2011-03-03 (Estimated); Last update posted 2014-04-28 (Estimated); Status verified 2014-04

CONDITIONS: Umbilical Hernia
Keywords: Umbilical Hernia Repair; PVP Mesh
MeSH Terms: conditions — Hernia, Umbilical

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Meshes-devices using dual-sided mesh technology have been developed for the specific indication of small ventral hernias. The design of these meshes allows introduction of a mesh of appropriate size to cover the hernia defect, through a small incision. This technique is very attractive for the surgeon and the patients because the mesh usually can be introduced through a nearly invisible scar in the umbilicus. The avoidance of fixation sutures omits the pain related to these sutures. Short-term results and patient satisfaction are very favorable, encouraging the surgeons to continue with the technique, although long-term results of these meshes in good quality studies are lacking.

DETAILED DESCRIPTION:
The aim of this study is to evaluate the safety and efficacy at 12 months after repair of small and medium ventral hernias using PVP™. All patients operated between March 2009 and February 2011 at the participating centers, will be evaluated and described. Patients will be evaluated by clinical investigation, questioning and ultrasound. The investigators' main focus will be the incidence of complications related to the use of the device, during the first year. Also the investigators look at recurrence rate at 12 months, occurrence of pain at 12 months and foreign body feeling. The trial can be seen as a quality control of a cohort of patients treated with an innovative mesh device. No sponsoring from the company J&J will be asked or accepted.

ELIGIBILITY:
Inclusion Criteria:

* All patients that were treated at the participating centres with a PVP™ for the repair of an umbilical hernia or another abdominal wall hernia before February 2011.

Exclusion Criteria:

* no informed consent from the patient.
* patients lost to follow up.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All patients that were treated at the participating centres with a PVP™ for the repair of an umbilical hernia or another abdominal wall hernia before February 2011, are eligible for the trial.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2010-08; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Hernia recurrence | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Jan Bontinck, Principal Investigator — Algemeen Ziekenhuis Maria Middelares
Locations (1):
- AZ Maria Middelares, Ghent, Oost Vlaanderen, Belgium

REFERENCES:
- [Result] Bontinck J, Kyle-Leinhase I, Pletinckx P, Vergucht V, Beckers R, Muysoms F. Single centre observational study to evaluate the safety and efficacy of the Proceed Ventral Patch to repair small ventral hernias. Hernia. 2014 Oct;18(5):671-80. doi: 10.1007/s10029-013-1140-5. Epub 2013 Jul 24. PMID 23881401